CLINICAL TRIAL: NCT02842281
Title: Intestinal Microbiome Fructan Metabolism and Symptom Generation in Childhood IBS
Brief Title: Microbiome Fructan Metabolism and Symptoms in Childhood IBS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Baylor College of Medicine (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, Bruno Chumpitazi, Assistant Professor, Baylor College of Medicine
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Other
Other Study IDs: H-34372; K23DK101688 (NIH)
Record Dates: First submitted 2016-07-15; First posted 2016-07-22 (Estimated); Last update posted 2021-01-22 (Actual); Status verified 2021-01

CONDITIONS: Irritable Bowel Syndrome (IBS)
MeSH Terms: conditions — Irritable Bowel Syndrome | interventions — Fructans; fructooligosaccharide; maltodextrin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Fructan (Active Comparator): Fructans will be provided for 72 hours.
  Interventions: Other: Fructan
- Maltodextrin (Placebo Comparator): Maltodextrin will be provided for 72 hours.
  Interventions: Other: Maltodextrin

INTERVENTIONS:
Other: Fructan — Short-chain oligosaccharide primarily composed of fructose polymers
  Other Names: fructo-oligosaccharides
  Arms: Fructan
Other: Maltodextrin — Polysaccharide produced from starch
  Arms: Maltodextrin

SUMMARY:
This study evaluates whether the gut microbiome is involved in determining whether children with irritable bowel syndrome (IBS) develop worsening GI symptoms (e.g. pain) when given fructans (a sugar often found in wheat). Participants will both receive a diet with fructans and a diet without fructans.

DETAILED DESCRIPTION:
Fructans (fructo-oligosaccharides) are a type of carbohydrate which can not be hydrolyzed by humans. It is commonly found in wheat in the American diet. After ingestion they arrive essentially intact into the colon where they are metabolized by the colonic microbiome. Fructan avoidance has been found to help decrease gastrointestinal symptoms (e.g. pain) in those with IBS.

However not all individuals with IBS have worsening symptoms when eating fructans in their diet. This study seeks to evaluate whether the microbiome is involved in determining whether an individual with IBS has worsening symptoms with fructan ingestion.

Following a one week baseline period, participants will be randomized in a double-blind cross-over fashion to either a 72 hour meal period with fructans or a 72 hour meal period with maltodextrin (placebo). A washout period of at least 10 days will occur in between. Symptoms will be captured using a stool and pain diary. Stool specimens and urine specimens will be obtained at baseline and during the dietary interventions. Breath hydrogen testing will be obtained during the dietary interventions.

ELIGIBILITY:
Inclusion Criteria:

* Children ages 7-17 years
* Children with IBS will meet Rome III criteria per the Rome III questionnaire
* Healthy children will not have chronic conditions
* English speaking and able to read/write in English

Exclusion Criteria:

* Previous bowel surgery
* Documented gastrointestinal disorder (e.g. ulcerative colitis)
* Serious chronic medical condition (e.g. diabetes)
* Weight and/or height are greater than or less than 2 standard deviations for age
* Chronic conditions with GI symptoms (e.g. cystic fibrosis)
* Antibiotics within the past 3 months
* Pregnancy
* Autism spectrum disorder and/or significant developmental delay
* Mood disorders (e.g. major depression)
* Known post-infectious etiology

Ages: 7 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 55 (Actual)
Dates: Start 2014-09; Primary Completion 2019-03 (Actual); Study Completion 2019-12 (Actual)

PRIMARY OUTCOMES:
Operational Taxonomic Units (microbiome composition derived from 16s rRNA sequencing) | Three days
  Children with IBS who have worsening GI symptoms with fructans vs. those who do not
Microbiome metabolic signatures related to fructan metabolism | Three days
  Children with IBS who have worsening GI symptoms with fructans vs. those who do not
Metabolic products of fructan metabolism | Three days
  In those with IBS who have worsening symptoms when given fructans, the investigators will correlate fructan metabolic byproducts with GI symptoms (e.g. pain)

SECONDARY OUTCOMES:
Microbiome related signatures | Three days
  Healthy children will have their microbiome signatures (composition, metabolic signatures related to fructan metabolism, and metabolic products of fructan metabolism) compared to children with IBS
Overall microbiome metabolic signatures | Three days
  Children with IBS who have worsening GI symptoms vs. those who do not
Overall metabolic products | Three days
  Following a fructan challenge in children with IBS who develop worsening GI symptoms vs. those who do not
Breath hydrogen and methane production symptoms | Three days
  Children with IBS who have worsening GI symptoms when given fructans vs. those who do not

CONTACTS AND LOCATIONS:
Overall Officials: Bruno Chumpitazi, MD, MPH, Principal Investigator — Assistant Professor
Locations (2):
- United States (2):
  - Children's Nutrition Research Center, Houston, Texas
  - Texas Children's Hospital, Houston, Texas

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Derived] Chumpitazi BP, McMeans AR, Vaughan A, Ali A, Orlando S, Elsaadi A, Shulman RJ. Fructans Exacerbate Symptoms in a Subset of Children With Irritable Bowel Syndrome. Clin Gastroenterol Hepatol. 2018 Feb;16(2):219-225.e1. doi: 10.1016/j.cgh.2017.09.043. Epub 2017 Sep 29. PMID 28970147